CLINICAL TRIAL: NCT01499056
Title: Evaluation the Side Effect of Bone Marrow Derived Mesenchymal Stem Cell in Patients With Osteoarthritis of Hip Joint
Brief Title: Mesenchymal Stem Cell Transplantation in Osteoarthritis of Hip Joint
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-008
Record Dates: First submitted 2011-12-17; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2010-01

CONDITIONS: Hip Osteoarthritis
Keywords: osteoarthritis; hip joint; mesenchymal stem cell
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hip osteoarthritis (Experimental): The patients with hip joint osteoarthritis who underwent cell injection
  Interventions: Biological: stem cell injection

INTERVENTIONS:
Biological: stem cell injection — intra articular inection of mesenchymal stem cell

SUMMARY:
Osteoarthritis of the hip is a common type of osteoarthritis which can cause significant problems. First-line of management for patient with osteoarthritis consists of weight reduction, education, and analgesic medication. If necessary, invasive treatment like total hip replacement are performed for the patient. The objective of this study was to assess the safety of bone marrow mesenchymal stem cells (BM-MSCs) implantation in patients with hip osteoarthritis

DETAILED DESCRIPTION:
This is a phase one clinical study designed to investigate the safety of intra-articular injection of cultured autologous BM-MSCs in patients with severe hip osteoarthritis candidate for total hip replacement. All subjects will undergo bone marrow aspiration. Autologous MSCs will be extracted and cultured for 4 weeks. Patients will receive intra-articular injection of cultured MSCs under the guide of fluoroscopy. Paraclinical studies (X-Ray and MRI) will be done before and 6 months after treatment. Pain relief and functional improvement of the joint will be assessed by VAS, WOMAC, and Harris Hip Score questionnaire before treatment, and 2 and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis diagnosed by MRI
* End stage osteoarthritis candidate for total hip replacement

Exclusion Criteria:

* Pregnancy or lactating
* Positive tests for HIV, HCV, HBV
* Active neurologic disorder
* End organ damage
* Uncontrolled endocrine disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
swelling of hip joint | 2 months
  Evaluatin the swelling of hip joint by physical examination after intra articular injection.
deterioration of joint function | 2 months
  Evaluation deterioration of joint function by physical examination after intra articular cell injection.
skin allergic reaction | 1 week
  Evaluation the skin allergic reaction like erythema,rash,swelling after intra articular cell injection.
Respiratory reaction | 1 week
  Evaluation the Respiratory reaction like dyspenea by physical examination after imtra articular cell injection.

SECONDARY OUTCOMES:
Quantitative changes in pain intensity | 2 months
  Evaluation Quantitative changes in pain intensity measured by Visual Analogue Scale after intra articular cell injection 2 months after cell transplantation in compare with base line (before injection)
physical function improvement | 2 months
  Evaluation the physical function improvement Measured by WOMAC osteoarthritis index and Harris Hip Score.
subchondral bone edema | 2 months
  Evaluation the subchondral bone edema by MRI
cartilage thickness | 2 months
  measuring the cartilage thickness after cell transplantation by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan Cell therapy Center; Mohsen Emadeddin, MD, Principal Investigator — scientist
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Emadedin M, Ghorbani Liastani M, Fazeli R, Mohseni F, Moghadasali R, Mardpour S, Hosseini SE, Niknejadi M, Moeininia F, Aghahossein Fanni A, Baghban Eslaminejhad R, Vosough Dizaji A, Labibzadeh N, Mirazimi Bafghi A, Baharvand H, Aghdami N. Long-Term Follow-up of Intra-articular Injection of Autologous Mesenchymal Stem Cells in Patients with Knee, Ankle, or Hip Osteoarthritis. Arch Iran Med. 2015 Jun;18(6):336-44. PMID 26058927